CLINICAL TRIAL: NCT06639360
Title: Effects of Transcranial Magnetic Stimulation After Endovascular Treatment for Acute Ischemic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY20242288-C-1
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Stroke, Acute; Endovascular Thrombectomy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active-cTBS group (Experimental): Patients assigned to the Active-cTBS group will be treated with cTBS and usual medical treatment after endovascular treatment
  Interventions: Device: Transcranial Magnetic Stimulation Active
- Sham-cTBS group (Sham Comparator): Patients assigned to the Sham-cTBS group will be treated with sham-cTBS and usual medical treatment after endovascular treatment
  Interventions: Device: Transcranial Magnetic Stimulation Sham

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation Active — The patients will be treated with cTBS and usual medical treatment after endovascular treatment
  Arms: Active-cTBS group
Device: Transcranial Magnetic Stimulation Sham — The patients will be treated with sham-cTBS and usual medical treatment after endovascular treatment
  Arms: Sham-cTBS group

SUMMARY:
This is a multicenter, randomized, double-blind, sham-controlled trial, to determine the efficacy and safety of cTBS in treating patients with acute ischemic stroke after endovascular treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute anterior circulation ischemic stroke aged between 18 and 80 years old.
2. Imaging suggests that the infarction is caused by occlusion of the terminal portion of the internal carotid artery or the M1/M2 segment of the middle cerebral artery.
3. A head CT within 24 hours of onset indicates an ASPECT score ≥6, and meets the guideline-recommended criteria for thrombectomy.
4. Pre-stroke mRS score is ≤1.
5. NIHSS score before thrombectomy is between 6 and 25.
6. With vascular recanalization of mTICI > 2b/3.
7. Informed consent form signed.

Exclusion Criteria:

1. Patients with contraindications to TMS treatment, such as those with metallic foreign objects in the head, pacemakers, implantable drug pumps, cochlear implants, etc.;
2. Patients with epilepsy, increased intracranial pressure, tumors, acute cerebral hemorrhage, or other severe neurological diseases, and those with severe functional impairment of organs such as the heart, liver, and kidneys;
3. Head CT/MRI indicates midline shift or significant mass effect, or patients planned for surgical intervention;
4. Head CT/MRI suggests acute cerebral infarction in both sides;
5. Patients who are pregnant or breastfeeding;
6. Patients with severe mental disorders or dementia who cannot cooperate with follow-up;
7. Patients with other severe diseases resulting in an expected survival of less than 90 days;
8. Patients who are participating in other interventional clinical studies within 30 days before the start of this study or after the onset of this condition;
9. Patients who cannot cooperate with informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-02 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of infarct volumes from baseline to Day 5 | 5 days after enrollment
Death | The first 5 days after enrollment
NIHSS at Day 5 | 5 days after enrollment

SECONDARY OUTCOMES:
Early neurological deterioration | 3 days after enrollment
  proportion of patients with an increase of ≥4 points in NIHSS at 3 days
Final infarct volume | 5 days after enrollment
  The infarct volume on DWI at 5 days
Intracranial hemorrhage incidence | 24h after enrollment
Proportion of patients with symptomatic intracranial hemorrhage | 90 days after enrollment
Proportion of patients with mRS 0-2 | 90 days after enrollment
Barthel Index score | 90 days after enrollment
Stroke recurrence | 90 days after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No